CLINICAL TRIAL: NCT05165914
Title: Midazolam Effect on Agitation Postnasal Surgery: A Double Blinded Randomized Controlled Trial
Brief Title: Midazolam Effect on Agitation Postnasal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordanian Royal Medical Services (Other)
Responsible Party: Principal Investigator, Ahmad Ben Tareef, Principal Investigator, Jordanian Royal Medical Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JordanianRoyalMS
Record Dates: First submitted 2021-12-03; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Agitation
Keywords: Agitation; Midazolam; Nasal surgery; Emergence
MeSH Terms: conditions — Psychomotor Agitation | interventions — Midazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam group (Active Comparator): In the midazolam group, patients double blindly received 0.03 mg.kg-1 midazolam intravenously just before emergence from general anesthesia.
  Interventions: Drug: Intravenous midazolam before emergence from general anesthesia
- Placebo group (Placebo Comparator): In the placebo group, patients double blindly received normal saline of similar volume to midazolam just before emergence from general anesthesia.
  Interventions: Drug: Intravenous normal saline before emergence from general anesthesia

INTERVENTIONS:
Drug: Intravenous midazolam before emergence from general anesthesia — Intravenous administration of 0.03 mg/kg midazolam just before emergence from anesthesia.
  Other Names: Versed
  Arms: Midazolam group
Drug: Intravenous normal saline before emergence from general anesthesia — Intravenous administration of normal saline just before emergence from anesthesia.
  Other Names: Normal saline 0.9%
  Arms: Placebo group

SUMMARY:
Postoperative agitation is a common complication, it's incidence post head and neck surgery is around 11-26%. Avoiding such complication is mandatory to facilitate patient's recovery and reduce risk of postoperative agitation related complications. Our study aims to detect the incidence of agitation following nasal surgery, and to determine the midazolam effect on agitation, when administered just before emergence from anesthesia.

DETAILED DESCRIPTION:
This is a prospective, single centre, double blinded randomized controlled trial, which was conducted from May 2021 to November 2021. An ethical approval was obtained from the local research ethical board in the Jordanian Royal Medical Services on May 26, 2021, in addition to an informed written consent from every patient. Subjects with American Society of Anesthesiologists (ASA) of either grade 1 or 2, aged from 16 to 59 years, undergoing nasal surgery such as; septoplasty (SP), open septorhinoplasty (OSRP) and functional endoscopic sinus surgery (FESS) were included in the study. A sample size of 100, 50 in each group was found to be enough to achieve the study purposes using G*Power computer program, considering alpha set at 0.05; medium effect size and study power 80%. Subjects were randomly assigned into two groups, midazolam group and placebo group. In the midazolam group, patients double blindly received 0.03 mg.kg-1 midazolam intravenously just before emergence from general anesthesia. On the other hand, placebo group's patients double blindly received normal saline of similar volume to midazolam just before emergence from general anesthesia. A computerized random number generator was utilized to provide the codes for midazolam and normal saline syringes. Patients otherwise received the same general anesthetic technique, including medications and equipments by the same anesthesiologist. The maximum Richmond Agitation Sedation Scale (RASS) score, from the time of extubation till patient's handover to postanesthesia care unit (PACU) was observed and documented by the same anesthesiologist and it was the basis for agitation diagnosis, therefore, the primary outcome was RASS score of +2 or more.

Anesthetic technique: No premedication was given to any patient. All patients received intravenous fentanyl 1.5 mcg.kg-1, propofol 2 mg.kg-1 and cisatracurium 0.2 mg.kg-1 for induction of general anesthesia. This was followed by manual ventilation for 4 minutes and intubation. Anesthesia was maintained by 1 MAC (Minimal Alveolar Concentration) of desflurane for all patients, in addition to remifentanil infusion (0.02 - 2.0 mcg.kg-1.minute-1) to aid analgesia and controlled hypotension with a mean arterial pressure not less than 60 mm Hg. An oropharyngeal pack was inserted for everyone and taken out gently before emergence and extubation. All patients received dexamethasone 8 mg, ondansetron 4 mg, 1 gram of paracetamol and 0.1 mg.kg-1 morphine intravenously. Morphine was given at the end of surgery by the time of turning the remifentanil infusion off. Midazolam or normal saline was randomly and blindly administered to patients using a 3 ml syringe (1mg.ml-1) at time of turning the remifentanil infusion off. By the end of surgery, desflurane was turned off and nobody received reversal for the cisatracurium, then smooth suctioning of the oral cavity was performed followed by awake extubation. No stimulation was used to aid patient's recovery except for gentle verbal commands.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) of either grade 1 or 2.
* Age from 16 to 59 years.
* Patients undergoing nasal surgery such as; septoplasty (SP), open septo-rhinoplasty (OSRP) and functional endoscopic sinus surgery (FESS).

Exclusion Criteria:

* ASA grade more than 2.
* Age less than 16 or more than 59 years.
* Any surgery that doesn't involve the nose or sinuses.

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Development of agitation | Up to one hour after extubation
  Agitation is diagnosed using the maximum score of Richmond Agitation Sedation Scale (RASS)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Ben Tareef, MD, Principal Investigator — Jordanian Royal Medical Services
Locations (1):
- Royal Medical Services, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim SY, Kim JM, Lee JH, Song BM, Koo BN. Efficacy of intraoperative dexmedetomidine infusion on emergence agitation and quality of recovery after nasal surgery. Br J Anaesth. 2013 Aug;111(2):222-8. doi: 10.1093/bja/aet056. Epub 2013 Mar 22. PMID 23524149
- [Result] Kim KM, Lee KH, Kim YH, Ko MJ, Jung JW, Kang E. Comparison of effects of intravenous midazolam and ketamine on emergence agitation in children: Randomized controlled trial. J Int Med Res. 2016 Apr;44(2):258-66. doi: 10.1177/0300060515621639. Epub 2016 Feb 15. PMID 26880794
- [Result] Cho EJ, Yoon SZ, Cho JE, Lee HW. Comparison of the effects of 0.03 and 0.05 mg/kg midazolam with placebo on prevention of emergence agitation in children having strabismus surgery. Anesthesiology. 2014 Jun;120(6):1354-61. doi: 10.1097/ALN.0000000000000181. PMID 24566243
- [Result] Sherwin TS, Green SM, Khan A, Chapman DS, Dannenberg B. Does adjunctive midazolam reduce recovery agitation after ketamine sedation for pediatric procedures? A randomized, double-blind, placebo-controlled trial. Ann Emerg Med. 2000 Mar;35(3):229-38. doi: 10.1016/s0196-0644(00)70073-4. PMID 10692189